CLINICAL TRIAL: NCT03696615
Title: Short Term Effects of Kettlebell Swings on Low Back Pain Pressure Threshold in Healthy Young Adults Utilizing a Tabata Protocol Format.
Brief Title: Kettlebell Swings & Low Back Pressure Pain Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 020551
Record Dates: First submitted 2016-05-10; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain
Keywords: high-intensity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tabata Kettlebell Swings (Experimental): Participants in this group performed:
  1. A brief dynamic warm-up (10 clockwise and counterclockwise arm circles, 10 horizontal arm swings, and 15 air squats)
  2. Receive instruction on the kettlebell swing
  3. Performed a high-intensity workout in a "Tabata Kettlebell Swings" format, which involves 20 seconds of all out effort followed by 10 seconds of rest, repeated for a total of 8 times.
  Interventions: Other: Tabata Kettlebell Swing Workout
- Control Group (Active Comparator): Participants in this group performed:
  1. A brief dynamic warm-up (10 clockwise and counterclockwise arm circles, 10 horizontal arm swings, and 15 air squats)
  Interventions: Other: Control

INTERVENTIONS:
Other: Tabata Kettlebell Swing Workout — See description of experimental arm.
  Arms: Tabata Kettlebell Swings
Other: Control — see description of control arm
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether a high intensity kettlebell workout, utilizing a Tabata protocol format, can decrease objective measures of pain pressure threshold in subjects without low back pain. The results of the study could have implications for the use of high intensity kettlebell workouts in the rehabilitation of patients with low back pain.

DETAILED DESCRIPTION:
The kettlebell swing is a full body, posterior-chain focused, ballistic exercise shown to register large recruitment of the gluteal muscles, which are frequently weak in a patients suffering from low back pain. The Tabata protocol is a high-intensity training protocol in which subjects perform 20 seconds of all out effort (i.e. as many swings as possible), followed by 10 seconds of rest, repeated for a total of eight rounds. The rapid contraction-relaxation cycles utilized in the kettlebell swing are theorized to aid in the pumping out of muscle metabolites in the low back musculature, thus providing potential relief of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Those subjects between the ages of 18 and 45
* No current low back pain or pre-existing injuries that may be currently affecting them
* No positive response on the Health History questionnaire and PAR-Q.

Exclusion Criteria:

* Current low back pain
* Pre-existing injuries currently affecting the subject
* Positive response on the Health History Questionnaire or PAR-Q
* We will also be excluding minors and prisoners from this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pressure measured in kilopascals | 1 minute post-intervention
  Pressure algometry measured in kilopascals

CONTACTS AND LOCATIONS:
Overall Officials: William J Hanney, PhD, Study Director — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States